CLINICAL TRIAL: NCT06257654
Title: One-year Results After Single-center Water Vapor Thermal Therapy for Symptomatic Benign Prostatic Hyperplasia.
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Ass. Prof., Hisar Intercontinental Hospital
Other Study IDs: 26.01.2024/24-2
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- singel
  Interventions: Device: REZUM

INTERVENTIONS:
Device: REZUM — The 3rd and 12th month follow-ups of the patients who underwent REZUM operation were evaluated.

SUMMARY:
Objective: Rezūm vapor ablation is a minimally invasive treatment for benign prostatic hyperplasia (BPH) that uses injections of sterile water vapor directly into the prostate for tissue ablation. Although Rezūm is currently indicated for use in men with prostate sizes ≥30 and ≤80 ml, it is unclear how effective Rezūm is for men in urinary retention. The investigators sought to determine whether Rezūm is effective in the treatment of catheter-dependent urinary retention secondary to BPH.

DETAILED DESCRIPTION:
The data of participants who underwent Rezūm operation with the diagnosis of BPH between 2021 and 2023 were evaluated retrospectively. The investigators evaluated procedure details and evaluated pre- and post-Rezūm (including International Prostate Symptom Score (IPSS), IPSS quality of life (IPSS-QOL), prostate volumes, maximum flow (Qmax), post-void residual urine volume, IEEF-5, ejaculation dysfunction). The investigators examined variables at 6 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

-Benign prostatic hyperplasia

Exclusion Criteria:

* Prostate cancer
* Parkinson's disease,
* Neurogenic bladder
* Overactive bladder
* Bladder calculus,
* Bladder Tumor
* Urinary infection
* Alzheimer's disease

Ages: 40 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male patients with prostate symptoms
Study Population: male patients with prostate symptoms
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score, | 1 years
  Scoring from 1-35, An increase in symptoms means an increase in the score, or a decrease in symptoms means a low score.
quality of life index | 1 years
  Scoring from 1-4, An increase in the quality of life means an increase in the score, or a decrease in the quality of life means a decrease in the score.
q max | 1 years
  ml/sn

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Basri Cakiroglu, Istanbul
  - Hisar Intercontinental Hospital, Istanbul